CLINICAL TRIAL: NCT02691637
Title: Effect of Helicobacter Pylori Eradication on the Reversibility of Atrophic Gastritis and Intestinal Metaplasia in Korean Patients.
Brief Title: Effect of H. Pylori Eradication on the Reversibility of Atrophic Gastritis and Intestinal Metaplasia in Korean Patients
Status: Completed | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: National Clinical Research Coordination Center, Seoul, Korea (Other Government)
Responsible Party: Principal Investigator, Nayoung Kim, Professor, Seoul National University Bundang Hospital
Other Study IDs: B-0602/030-001
Record Dates: First submitted 2016-02-14; First posted 2016-02-25 (Estimated); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Helicobacter Pylori Infection; Atrophic Gastritis; Intestinal Metaplasia
Keywords: Helicobacter pylori infection; Eradication treatment; Reversibility; atrophic gastritis; intestinal metaplasia
MeSH Terms: conditions — Gastritis, Atrophic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- H. pylori eradication group: Patients who have had H. pylori infection. After diagnosis of H. pylori infection, the patients who subsequently received successful H. pylori eradication treatment according to appropriate indication.
- Control Group: Patients who still have H. pylori infection. The patients of control group do not have successful H. pylori eradication result or do not received eradication treatment for any reason.

SUMMARY:
Helicobacter pylori (H. pylori) infection has been associated with a development of atrophic gastritis and intestinal metaplasia. H. pylori related atrophic gastritis and intestinal metaplasia have been regarded as pre-malignant lesion. However, the role of H. pylori eradication treatment in the reversibility of atrophic gastritis and intestinal metaplasia has not been clearly defined. The aim of the present study was to investigate the relationship between H. pylori eradication and the reversibility of atrophic gastritis and intestinal metaplasia in Korean patients.

DETAILED DESCRIPTION:
It is a prospective, case-control study to compare the status of atrophic gastritis and intestinal metaplasia from the patients who undergo H. pylori eradication treatment or not. After enrollment, each patient will be receive annual surveillance upper gastrointestinal endoscopy. The present investigators will monitor the status of atrophic gastritis and intestinal metaplasia annually and finally compare the reversibility of them.

ELIGIBILITY:
Inclusion Criteria:

- Patients who diagnosis of H. pylori infection

* Patients presenting with H. pylori related gastrointestinal disease and/or
* Patients do not have H. pylori related gastrointestinal disease. But, want H. pylori eradication

Exclusion Criteria:

- Age under 18 years Previous eradication treatment for H. pylori Patients who took any drug which could influence the study results such as proton pump inhibitor, antibiotics within 4 weeks History of gastrectomy Advanced gastric cancer or other malignancy Abnormal liver function or liver cirrhosis Abnormal renal function or chronic kidney disease Other severe concurrent diseases Previous allergic reactions to the study drugs Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have H. pylori related gastrointestinal disease and/or Patients who do not have H. pylori related gastrointestinal disease. But, want H. pylori eradication
Sampling Method: Probability Sample
Enrollment: 1450 (Actual)
Dates: Start 2006-02; Primary Completion 2022-01 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
The improvement of Atrophic Gastritis and Intestinal metaplasia score | per 1 year
  The improvement of Atrophic Gastritis and Intestinal metaplasia was defined as improvement of score compared with baseline.
  The histological features of the gastric mucosa were recorded using updated Sydney system scores, that is, 0 = none, 1 = mild, 2 = moderate, and 3 = marked.(Am J Surg Pathol 1996;20:1161-81.) Outcome measure will be done annually (per 1 year), final follow-up is 2019

CONTACTS AND LOCATIONS:
Overall Officials: Officials Officials, Officials, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No